CLINICAL TRIAL: NCT03945409
Title: Validation of a New Automated System for Continuous Real-time Monitoring of Transpulmonary Pressure During Invasive Mechanical Ventilation in Patients With Acute Respiratory Failure
Brief Title: New Automated System for Continuous Real-time Monitoring of Transpulmonary Pressure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Davide Chiumello, Professor, University of Milan
Other Study IDs: INNOVENT-2019
Record Dates: First submitted 2019-04-17; First posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Acute Respiratory Failure; Ventilator-Induced Lung Injury
Keywords: ARDS; Respiratory Mechanics; Transpulmonary pressure; Pleural pressure
MeSH Terms: conditions — Ventilator-Induced Lung Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: OPTIVENT — OPTIVENT (SIDAM SRL, Mirandola, Italy) is a new fully automated and self-calibrating system that allows a real-time monitoring and recording of airway pressure and esophageal pressure during mechanical ventilation. The system required the insertion of an esophageal balloon catheter and an airway pressure transducer.

SUMMARY:
Patients admitted to Intensive Care Unit often are affected by acute respiratory failure at admission or during hospital stay, with a mortality of 30%.

Treatment remains largely supportive with mechanical ventilation as the mainstay of management by improving the hypoxemia and reducing the work of breathing; however, the mechanical forces generated during ventilation can further enhance pulmonary inflammation and edema, a process that has been termed ventilator induced lung injury (VILI). Consequently, in clinical practice the lung protective ventilation is mainly based on the reduction of the tidal volume, the airway and the transpulmonary plateau pressure. A good clinical practice is based on the assessment of changes in respiratory mechanics.

Aim of the study is to determine the accuracy of the OPTIVENT system in measuring transpulmonary pressure, comparing it with the systems currently in use in our Operative Unit.

ELIGIBILITY:
Inclusion Criteria:

* acute respiratory failure
* invasive mechanical ventilation.

Exclusion Criteria:

* haemodynamic instability
* presence of barotrauma
* esophageal disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients admitted to our Intensive Care Unit affected by acute respiratory failure, mechanically ventilated.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-03-28 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Measure of transpulmonary pressure (cmH2O). | Day 1.
  Validation of the new system in terms of accuracy and precision. The accuracy of the OPTIVENT system in measuring transpulmonary pressure, comparing it with the systems currently in use, will be assessed by measure of airway and esophageal pressure at the end of an inspiratory and expiratory hold.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - ASST-Santi Paolo e Carlo, San Paolo Hospital, Milan, MI
  - Ospedale San Paolo - Polo Universitario, ASST Santi Paolo e Carlo, Milan, MI

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Mac Sweeney R, McAuley DF, Matthay MA. Acute lung failure. Semin Respir Crit Care Med. 2011 Oct;32(5):607-25. doi: 10.1055/s-0031-1287870. Epub 2011 Oct 11. PMID 21989697
- [Background] Vincent JL, de Mendonca A, Cantraine F, Moreno R, Takala J, Suter PM, Sprung CL, Colardyn F, Blecher S. Use of the SOFA score to assess the incidence of organ dysfunction/failure in intensive care units: results of a multicenter, prospective study. Working group on "sepsis-related problems" of the European Society of Intensive Care Medicine. Crit Care Med. 1998 Nov;26(11):1793-800. doi: 10.1097/00003246-199811000-00016. PMID 9824069
- [Background] Vincent JL, Akca S, De Mendonca A, Haji-Michael P, Sprung C, Moreno R, Antonelli M, Suter PM; SOFA Working Group. Sequntial organ failure assessment. The epidemiology of acute respiratory failure in critically ill patients(*). Chest. 2002 May;121(5):1602-9. doi: 10.1378/chest.121.5.1602. PMID 12006450
- [Background] Slutsky AS, Ranieri VM. Ventilator-induced lung injury. N Engl J Med. 2013 Nov 28;369(22):2126-36. doi: 10.1056/NEJMra1208707. No abstract available. PMID 24283226
- [Background] Dreyfuss D, Saumon G. Ventilator-induced lung injury: lessons from experimental studies. Am J Respir Crit Care Med. 1998 Jan;157(1):294-323. doi: 10.1164/ajrccm.157.1.9604014. No abstract available. PMID 9445314
- [Background] Gattinoni L, Carlesso E, Cadringher P, Valenza F, Vagginelli F, Chiumello D. Physical and biological triggers of ventilator-induced lung injury and its prevention. Eur Respir J Suppl. 2003 Nov;47:15s-25s. doi: 10.1183/09031936.03.00021303. PMID 14621113
- [Background] Tremblay L, Valenza F, Ribeiro SP, Li J, Slutsky AS. Injurious ventilatory strategies increase cytokines and c-fos m-RNA expression in an isolated rat lung model. J Clin Invest. 1997 Mar 1;99(5):944-52. doi: 10.1172/JCI119259. PMID 9062352
- [Background] Akoumianaki E, Maggiore SM, Valenza F, Bellani G, Jubran A, Loring SH, Pelosi P, Talmor D, Grasso S, Chiumello D, Guerin C, Patroniti N, Ranieri VM, Gattinoni L, Nava S, Terragni PP, Pesenti A, Tobin M, Mancebo J, Brochard L; PLUG Working Group (Acute Respiratory Failure Section of the European Society of Intensive Care Medicine). The application of esophageal pressure measurement in patients with respiratory failure. Am J Respir Crit Care Med. 2014 Mar 1;189(5):520-31. doi: 10.1164/rccm.201312-2193CI. PMID 24467647